CLINICAL TRIAL: NCT03232216
Title: Vitamin D Supplementation in Patients With Operated Tibia Fracture and Low Vitamin D. Does it Improve Healing Rate?. Randomized Controlled Trial
Brief Title: Vitamin D Supplementation and Tibia Fracture. Does it Improve Healing Rate?
Acronym: ViDco
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital del Trabajador de Santiago (Other)
Responsible Party: Principal Investigator, Sebastián Drago Pérez, Orthopedic Surgeon, Hospital del Trabajador de Santiago
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ViDco
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Tibial Fractures; Vitamin D Deficiency; Fracture Healing
MeSH Terms: conditions — Tibial Fractures; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vitamin D3 supplementation. Deficiency. (Experimental): Vitamin D3 50.000 UI in each packet of powder for solution. Two packets every week for 5 weeks.
  Interventions: Dietary Supplement: Vitamin D3.
- Placebo. Deficiency. (Placebo Comparator): Placebo of Vitamin D3 50.000 UI in each packet of powder for oral solution. Two packets every week for 5 weeks.
  Interventions: Dietary Supplement: Placebo
- Vitamin D3 supplementation.Insufficiency (Experimental): Vitamin D3 50.000 UI in each packet of powder for oral solution. Two packets every week for 3 weeks.
  Interventions: Dietary Supplement: Vitamin D3.
- Placebo. Insufficiency. (Placebo Comparator): Placebo of Vitamin D3 50.000 UI in each packet of powder for oral solution. Two packets every week for 3 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3. — Vitamin D3 50.000 UI in each packet of powder for oral solution.
  Other Names: Cholecalciferol
  Arms: Vitamin D3 supplementation. Deficiency.; Vitamin D3 supplementation.Insufficiency
Dietary Supplement: Placebo — Placebo of Vitamin D3 50.000 UI in each packet of powder for oral solution.
  Arms: Placebo. Deficiency.; Placebo. Insufficiency.

SUMMARY:
This study evaluates the effect of Vitamin D3 supplementation in healing rate of tibia fractures in adult patients with low vitamin D. Half of participants will receive Vitamin D3 supplementation while the other will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* Tibial fracture
* ASA physical status classification system I-II.
* 25 hydroxyvitamin D below 30ng/ml)
* Fracture treatment with reamed intramedullary nail

Exclusion Criteria:

* Open Fractures Gustillo III B and III C
* Closed Soft tissue injury with Tscherne classification of III
* Acute Compartment Syndrome
* Pathology fractures (That occur in abnormal bone, for example in the presence of tumor, cyst or Paget disease)
* Other Fractures in lower limbs or spine that does not allow full weight bearing of the operated tibia after 4 weeks
* More than 7 days of evolution from fracture occurrence
* Diabetes mellitus with HbA1c more or equal than 7%
* Peripheral vascular disease
* Rickets
* Pre-existing disorders of the metabolism of Vitamin D and/or homeostasis of calcium and phosphorous (ie. Hepatic insufficiency, congenital defects of the vitamin D metabolism, disorders of the parathyroid glands, hypo or hyper calcemia)
* Renal failure with glomerular filtration rate below 60ml/min according to MDRD-4.
* Patients using nephrotoxic medications in high doses, requiring periodical monitoring of glomerular filtration rate
* Patients undergoing with nephrotic syndrome or that suffered it in the past
* Patients that suffered nephrolithiasis or urolithiasis
* Pregnant women
* Patients with allergy to vitamin D or other contraindications for vitamin D3 prescription
* Patients that are taking multivitamin supplements containing vitamin D and will not suspend taking them during the study.
* Patients that are not able to swallow a cup of water

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 682 (Estimated)
Dates: Start 2017-11-21 (Actual); Primary Completion 2021-08-18 (Estimated); Study Completion 2023-08-18 (Estimated)

PRIMARY OUTCOMES:
Fracture non union | 2 years
  Rate of fracture non union in each group

SECONDARY OUTCOMES:
Prevalence of low vitamin D in adults with tibia fracture | 10 days
  Using the first measurement of 25 hydroxyvitamin D
Time of fracture healing | 2 years
  Time that lasted consolidation, from surgery
Short Form 36 score (SF-36) | 2 years
  Health associated quality of life
EuroQol five dimensions questionnaire (EQ-5D) | 2 years
  Generic health status measurement
Knee Range of movement | 2 years
  Knee flexion and extension in degrees
Ankle Range of movement | 2 years
  Ankle flexion and extension in degrees
Superficial Infections | 2 years
  Incidence of superficial infections in each group
Deep infections | 2 years
  Incidence of superficial infections in each group
Visual Analogue Scale (VAS) | 2 years
  Pain measurement using VAS

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Drago, Principal Investigator — Hospital del Trabajador de Santiago
Locations (1):
- Hospital del Trabajador de Santiago, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manson JE, Brannon PM, Rosen CJ, Taylor CL. Vitamin D Deficiency - Is There Really a Pandemic? N Engl J Med. 2016 Nov 10;375(19):1817-1820. doi: 10.1056/NEJMp1608005. No abstract available. PMID 27959647
- [Background] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368
- [Background] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462
- [Background] Schwartz JB, Kane L, Bikle D. Response of Vitamin D Concentration to Vitamin D3 Administration in Older Adults without Sun Exposure: A Randomized Double-Blind Trial. J Am Geriatr Soc. 2016 Jan;64(1):65-72. doi: 10.1111/jgs.13774. PMID 26782853
- [Background] Talib HJ, Ponnapakkam T, Gensure R, Cohen HW, Coupey SM. Treatment of Vitamin D Deficiency in Predominantly Hispanic and Black Adolescents: A Randomized Clinical Trial. J Pediatr. 2016 Mar;170:266-72.e1. doi: 10.1016/j.jpeds.2015.11.025. Epub 2015 Dec 18. PMID 26707619
- [Background] Vieth, R: The pharmacology of vitamin D. Vitam D 2011;1041-1066. doi:10.1016/B978-0-12-381978-9.10057-5
- [Background] Antonova E, Le TK, Burge R, Mershon J. Tibia shaft fractures: costly burden of nonunions. BMC Musculoskelet Disord. 2013 Jan 26;14:42. doi: 10.1186/1471-2474-14-42. PMID 23351958
- [Background] Khaw KT, Stewart AW, Waayer D, Lawes CMM, Toop L, Camargo CA Jr, Scragg R. Effect of monthly high-dose vitamin D supplementation on falls and non-vertebral fractures: secondary and post-hoc outcomes from the randomised, double-blind, placebo-controlled ViDA trial. Lancet Diabetes Endocrinol. 2017 Jun;5(6):438-447. doi: 10.1016/S2213-8587(17)30103-1. Epub 2017 Apr 28. PMID 28461159
- [Result] Sprague S, Petrisor B, Scott T, Devji T, Phillips M, Spurr H, Bhandari M, Slobogean GP. What Is the Role of Vitamin D Supplementation in Acute Fracture Patients? A Systematic Review and Meta-Analysis of the Prevalence of Hypovitaminosis D and Supplementation Efficacy. J Orthop Trauma. 2016 Feb;30(2):53-63. doi: 10.1097/BOT.0000000000000455. PMID 26429406
- [Result] Carrasco G M, Dominguez De L A, Martinez F G, Ihle S S, Rojas A V, Foradori C A, Marin L PP. [Vitamin D levels in older healthy Chilean adults and their association with functional performance]. Rev Med Chil. 2014 Nov;142(11):1385-91. doi: 10.4067/S0034-98872014001100004. Spanish. PMID 25694283
- [Result] Schweitzer D, Amenabar PP, Botello E, Lopez M, Saavedra Y, Klaber I. [Vitamin D levels among Chilean older subjects with low energy hip fracture]. Rev Med Chil. 2016 Feb;144(2):175-80. doi: 10.4067/S0034-98872016000200005. Spanish. PMID 27092671
- [Result] Souberbielle JC, Massart C, Brailly-Tabard S, Cavalier E, Chanson P. Prevalence and determinants of vitamin D deficiency in healthy French adults: the VARIETE study. Endocrine. 2016 Aug;53(2):543-50. doi: 10.1007/s12020-016-0960-3. Epub 2016 Apr 22. PMID 27106800
- [Result] Yu S, Fang H, Han J, Cheng X, Xia L, Li S, Liu M, Tao Z, Wang L, Hou L, Qin X, Li P, Zhang R, Su W, Qiu L. The high prevalence of hypovitaminosis D in China: a multicenter vitamin D status survey. Medicine (Baltimore). 2015 Feb;94(8):e585. doi: 10.1097/MD.0000000000000585. PMID 25715263
- [Result] Bodendorfer BM, Cook JL, Robertson DS, Della Rocca GJ, Volgas DA, Stannard JP, Crist BD. Do 25-Hydroxyvitamin D Levels Correlate With Fracture Complications? J Orthop Trauma. 2016 Sep;30(9):e312-7. doi: 10.1097/BOT.0000000000000639. PMID 27253482
- [Result] Bell A, Templeman D, Weinlein JC. Nonunion of the Femur and Tibia: An Update. Orthop Clin North Am. 2016 Apr;47(2):365-75. doi: 10.1016/j.ocl.2015.09.010. PMID 26772945
- [Result] Duan X, Al-Qwbani M, Zeng Y, Zhang W, Xiang Z. Intramedullary nailing for tibial shaft fractures in adults. Cochrane Database Syst Rev. 2012 Jan 18;1(1):CD008241. doi: 10.1002/14651858.CD008241.pub2. PMID 22258982